CLINICAL TRIAL: NCT03994211
Title: A Phase 1, Open-label, Parallel-group, Fixed-sequence Study to Investigate the Effect of the CYP3A Inducer Rifampin and the CYP3A Inhibitor Itraconazole on the Pharmacokinetics of Pamiparib (BGB-290) in Cancer Patients
Brief Title: Study to Investigate the Effect of Rifampin and Itraconazole on the Action of Pamiparib in Participants With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BGB-290-105; 2019-000112-28 (EudraCT Number)
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Results first posted 2023-05-23 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — pamiparib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (core phase) (Experimental): 60 mg pamiparib administered orally on Days 1 and 10 fasting 8 hours pre-dose 600 mg rifampin once a day from days 3 to 11 in the fasted state (at least 2 hours predose)
  Interventions: Drug: pamiparib 60 mg; Drug: rifampin
- Part B (core phase) (Experimental): Single dose of 20 mg pamiparib orally in the fasted state (at least 8 hours predose) on days 1 and 7 200 mg itraconazole once a day approximately 30 minutes after completing a meal Day 3 to day 8
  Interventions: Drug: pamiparib 20 mg; Drug: itraconazole
- Extension phase (Experimental): 60 mg pamiparib orally twice a day in 28-day cycles until progression of disease
  Interventions: Drug: pamiparib

INTERVENTIONS:
Drug: pamiparib 60 mg — Single dose of 60 mg pamiparib orally on Days 1 and 10
  Arms: Part A (core phase)
Drug: pamiparib 20 mg — Single dose of 20 mg pamiparib orally on days 1 and 7
  Arms: Part B (core phase)
Drug: itraconazole — 200 mg itraconazole once a day al Day 3 to day 8
  Arms: Part B (core phase)
Drug: rifampin — 600 mg rifampin once a day from days 3 to 11
  Arms: Part A (core phase)
Drug: pamiparib — 60 mg pamiparib orally twice a day in 28-day cycles
  Arms: Extension phase

SUMMARY:
The study was an open-label, parallel-group, fixed-sequence study in male and female cancer patients. The study consists of 2 phases: the Core Phase, which is divided into Part A and Part B, and the Extension Phase. Part A investigated the effect of CYP3A induction by rifampin on the single dose pharmacokinetics (PK) of pamiparib, and Part B investigated the effect of CYP3A inhibition by itraconazole on the single dose PK of pamiparib. Participants were offered participation in the Extension Phase, in which they received pamiparib until progression of disease, unacceptable toxicity, withdrawal of consent, or any other reason for discontinuation.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically confirmed advanced or metastatic solid tumors that are refractory or resistant to standard therapy or for which no suitable effective standard therapy exists.
3. Disease that is evaluable per RECIST Version 1.1 or Prostate Cancer Working Group-3 (PCWG-3)
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
5. Life expectancy ≥ 12 weeks
6. Adequate hematologic and end-organ function

Key Exclusion Criteria:

1. History of hypersensitivity to rifampin, any rifamycin or any of the components of the rifampin capsule (Part A).
2. History of hypersensitivity to itraconazole or any of the components of the itraconazole capsule (Part B).
3. Prior treatment with a poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor at therapeutic doses is allowed, provided that such treatment was not the most recent therapy (PARP inhibitor must have been discontinued ≥ 3 months prior to the first dose of pamiparib):

   - Participants who experienced prior severe toxicity to PARP inhibitors that in the opinion of the investigator precludes further treatment with PARP inhibitors should be excluded
4. Diagnosis of Myelodysplastic syndrome (MDS)
5. Active infection requiring systemic treatment
6. Any of the following cardiovascular criteria:

   1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before Day 1 of pamiparib administration
   2. Symptomatic pulmonary embolism ≤ 28 days before Day 1 of pamiparib administration
   3. Any history of acute myocardial infarction ≤ 6 months before Day 1 of pamiparib administration
   4. Any history of heart failure meeting New York Heart Association Classification III or IV ≤ 6 months before Day 1 of pamiparib

      - Participants with congestive heart failure or history of heart failure should be excluded from Part B (itraconazole)
   5. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before Day 1 of pamiparib administration
   6. Any history of cerebral vascular accident ≤ 6 months before Day 1 of pamiparib administration
7. Previous complete gastric resection or lap-band surgery, chronic diarrhea, active inflammatory gastrointestinal disease, known diverticular disease or any other disease-causing malabsorption syndrome

   - Gastroesophageal reflux disease under treatment with proton pump inhibitors is allowed
8. Active bleeding disorder, including gastrointestinal bleeding, as evidenced by hematemesis, significant hemoptysis, or melena ≤ 6 months before Day 1 of pamiparib administration
9. Use or anticipated need for food or drugs known to be strong or moderate CYP3A inhibitors or strong CYP3A inducers ≤ 14 days (or ≤ 5 half-lives if half-life is known) prior to Day 1 of pamiparib administration
10. Known history of intolerance to the excipients of the pamiparib capsule
11. Have known hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (4):
- Arensia Exploratory Medicine Llc, Tbilisi, Georgia
- Republican Clinical Hospital, Oncology Department, Chiinu, Moldova
- Szpital Luxmed, Warsaw, Poland
- Summit Clinical Research, Sro, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Mu S, Lin C, Skrzypczyk-Ostaszewicz A, Bulat I, Maglakelidze M, Skarbova V, Andreu-Vieyra C, Sahasranaman S. The pharmacokinetics of pamiparib in the presence of a strong CYP3A inhibitor (itraconazole) and strong CYP3A inducer (rifampin) in patients with solid tumors: an open-label, parallel-group phase 1 study. Cancer Chemother Pharmacol. 2021 Jul;88(1):81-88. doi: 10.1007/s00280-021-04253-x. Epub 2021 Mar 27. PMID 33772633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of a core phase and an extension phase. A total of 25 participants were enrolled in Poland, Moldova, Slovakia, and Georgia.
Pre-assignment Details: The screening period consisted of Days -28 to -1.
Groups:
- Core Phase: Arm A: Pamiparib + Rifampin: Participants received 60 milligrams (mg) pamiparib orally on Days 1 and 10 fasting 8 hours pre-dose + 600 mg rifampin orally from Day 3 to Day 11 fasting at least 2 hours pre-dose
- Core Phase: Arm B: Pamiparib + Itraconazole: Participants received 20 mg pamiparib orally on Days 1 and 7 fasting at least 8 hours pre-dose + 200 mg itraconazole orally 30 minutes after meal Day 3 to Day 8
- Extension Phase: Participants received 60 mg pamiparib orally twice a day in 28-day cycles until progression of disease, unacceptable toxicity, withdrawal of consent, or any other reason for discontinuation
Period: Core Phase
Arm/Group | Core Phase: Arm A: Pamiparib + Rifampin | Core Phase: Arm B: Pamiparib + Itraconazole | Extension Phase
Started | 12 | 13 | 0
Completed | 12 | 12 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Extension Phase
Arm/Group | Core Phase: Arm A: Pamiparib + Rifampin | Core Phase: Arm B: Pamiparib + Itraconazole | Extension Phase
Started | 0 | 0 | 24
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 24
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 20
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of pamiparib
Groups:
- Core Phase: Arm A: Pamiparib + Rifampin: Participants received 60 mg pamiparib orally on Days 1 and 10 fasting 8 hours pre-dose + 600 mg rifampin orally from Day 3 to Day 11 fasting at least 2 hours pre-dose
- Total: Total of all reporting groups
Arm/Group | Core Phase: Arm A: Pamiparib + Rifampin | Core Phase: Arm B: Pamiparib + Itraconazole | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.73) | 62.6 (12.96) | 60.7 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Pamiparib in Plasma for Part A
Time Frame: Part A: from Day -1 (admission) to Day 12 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12, 24, and 48 hours post-dose
Population: The pharmacokinetic (PK) population includes all participants who received at least 1 dose of pamiparib and have evaluable PK data. A participant was to be excluded from the PK summary statistics and statistical analysis if the participant had an adverse event (AE) of vomiting that occurred at or before 2 x median tmax.
Measure: Median (Full Range); unit: ng/mL
Groups:
- Part A: Pamiparib: Participants received 60 mg pamiparib orally on Days 1 and 10 fasting 8 hours pre-dose
- Part A: Pamiparib + Rifampin: Participants received 60 mg pamiparib Days 1 and 10 + 600 mg rifampin orally from Day 3 to Day 11 fasting at least 2 hours pre-dose
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 11 | 11
ng/mL | 1970 [1060.0 to 2700.0] | 1820 [1170.0 to 2500.0]
Statistical Analysis 1: Comparison: Part A: Pamiparib vs Part A: Pamiparib + Rifampin; Test type: Other; Geometric Mean Ratio Estimate = 0.94, 90% CI 2-sided [0.83 to 1.06]

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Pamiparib in Plasma for Part B
Time Frame: Part B: from Day -1 (admission) to Day 9 (discharge; ) 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12, 24, and 48 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Groups:
- Part B: Pamiparib: Participants received 20 mg pamiparib orally from Days 1 and 7 fasting at least 8 hours pre-dose
- Part B: Pamiparib + Itraconazole: Participants received pamiparib 20 mg fasting on Days 1 and 7 + 200 mg itraconazole orally 30 minutes after meal Day 3 to Day 8
Arm/Group | Part B: Pamiparib | Part B: Pamiparib + Itraconazole
Number analyzed (Participants) | 12 | 12
ng/mL | 730.5 [374.0 to 1130.0] | 752.5 [302.0 to 1130.0]
Statistical Analysis 1: Comparison: Part B: Pamiparib vs Part B: Pamiparib + Itraconazole; Test type: Other; Geometric Mean Ratio = 1.05, 90% CI 2-sided [0.95 to 1.15]

3. Primary Outcome: AUC From Time Zero to Time of Last Quantifiable Concentration Post-dose (AUC0-tlast) in Plasma for Part A
Time Frame: as for outcome 1
Population: The PK population includes all participants who received at least 1 dose of pamiparib and have evaluable PK data. A participant was to be excluded from the PK summary statistics and statistical analysis if the participant had an AE of vomiting that occurred at or before 2 x median tmax.
Measure: Median (Full Range); unit: hours*nanograms/milliLiter (h*ng/mL)
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 11 | 11
hours*nanograms/milliLiter (h*ng/mL) | 28868 [14680.8 to 46910.6] | 18351 [11097.3 to 24186.8]
Statistical Analysis 1: Comparison: Part A: Pamiparib vs Part A: Pamiparib + Rifampin; Test type: Other; Geometric Mean Ratio = 0.62, 90% CI 2-sided [0.54 to 0.70]

4. Primary Outcome: AUC From Time Zero to Time of Last Quantifiable Concentration Post-dose (AUC0-tlast) in Plasma for Part B
Time Frame: Part B: from Day -1 (admission) to Day 9 (discharge) 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12, 24, and 48 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours*nanograms/milliLiter (h*ng/mL)
Arm/Group | Part B: Pamiparib | Part B: Pamiparib + Itraconazole
Number analyzed (Participants) | 12 | 12
hours*nanograms/milliLiter (h*ng/mL) | 9163 [1797.5 to 20891.1] | 8894 [1528.1 to 19356.9]
Statistical Analysis 1: Comparison: Part B: Pamiparib vs Part B: Pamiparib + Itraconazole; Test type: Other; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.91 to 1.09]

5. Primary Outcome: AUC From Zero to Infinity (AUC0-inf) of Pamiparib in Plasma for Part A
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 9 | 11
hr*ng/mL | 28142 [14776 to 51942] | 18563 [11183 to 25615]
Statistical Analysis 1: Comparison: Part A: Pamiparib vs Part A: Pamiparib + Rifampin; Test type: Other; Geometric Mean Ratio = 0.57, 90% CI 2-sided [0.48 to 0.69]

6. Primary Outcome: AUC From Zero to Infinity (AUC0-inf) of Pamiparib in Plasma for Part B
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: hr*ng/mL
Groups:
- Part B:Pamiparib + Itraconazole: Participants received pamiparib 20 mg fasting on Days 1 and 7 + 200 mg itraconazole orally 30 minutes after meal Day 3 to Day 8
Arm/Group | Part B: Pamiparib | Part B:Pamiparib + Itraconazole
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 10072 [1828.4 to 25529.9] | 9353 [1541.9 to 23171.0]
Statistical Analysis 1: Comparison: Part B: Pamiparib vs Part B:Pamiparib + Itraconazole; Test type: Other; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.90 to 1.09]

7. Primary Outcome: AUC From Zero to 12 Hours (AUC0-12) of Pamiparib in Plasma for Part A
Time Frame: Part A: from Day -1 (admission) to Day 12 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, and 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 11 | 11
hr*ng/mL | 14642.90 [9502.6 to 20992.6] | 12262.61 [7908.4 to 15230.0]

8. Primary Outcome: AUC From Zero to 12 Hours (AUC0-12) of Pamiparib in Plasma for Part B
Time Frame: Part B: from Day -1 (admission) to Day 9 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, and 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Part B: Pamiparib | Part B: Pamiparib + Itraconazole
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 5097.06 [1640.4 to 8313.2] | 4647.47 [1413.5 to 8879.2]

9. Primary Outcome: AUC From Zero to 9 Hours (AUC0-9) of Pamiparib in Plasma for Part A
Time Frame: Part A: from Day -1 (admission) to Day 12 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, and 9 hours post-dose
Population: The PK population includes all participants who received at least 1 dose of pamiparib and have evaluable PK data. A participant was excluded from the PK summary statistics and statistical analysis if the participant had an AE of vomiting that occurred at or before 2 x median tmax.
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 11 | 11
hr*ng/mL | 11821.06 [7678.6 to 16561.4] | 10515.14 [6888.8 to 12813.6]

10. Primary Outcome: AUC From Zero to 9 Hours (AUC0-9) of Pamiparib in Plasma for Part B
Time Frame: Part B: from Day -1 (admission) to Day 9 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, and 9 hours post-dose
Population: as for outcome 9
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Part B: Pamiparib | Part B:Pamiparib + Itraconazole
Number analyzed (Participants) | 12 | 12
hr*ng/mL | 4267.86 [1525.3 to 6350.2] | 3812.39 [1315.8 to 7325.8]

11. Primary Outcome: Time of the Maximum Observed Concentration (Tmax) of Pamiparib for Part A
Time Frame: Part A: from Day -1 (admission) to Day 12 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 11 | 11
hours | 2.000 [1.00 to 4.00] | 2.000 [1.00 to 4.05]

12. Primary Outcome: Time of the Maximum Observed Concentration (Tmax) of Pamiparib for Part B
Time Frame: Part B: from Day -1 (admission) to Day 9 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Part B: Pamiparib | Part B:Pamiparib + Itraconazole
Number analyzed (Participants) | 12 | 12
hours | 2.000 [0.98 to 4.02] | 1.000 [0.95 to 2.02]

13. Primary Outcome: Apparent Terminal Elimination Half-life (t1/2) of Pamiparib in Plasma for Part A
Time Frame: Part A: from Day -1 (admission) to Day 12 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 9 | 11
hours | 13.381 [6.77 to 20.01] | 7.667 [5.09 to 11.39]

14. Primary Outcome: Apparent Terminal Elimination Half-life (t1/2) of Pamiparib in Plasma for Part B
Time Frame: Part B: from Day -1 (admission) to Day 9 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Part B: Pamiparib | Part B:Pamiparib + Itraconazole
Number analyzed (Participants) | 12 | 12
hours | 9.290 [4.48 to 19.14] | 11.179 [3.69 to 19.44]

15. Primary Outcome: Apparent Oral Clearance (CL/F) of Pamiparib in Plasma for Part A
Time Frame: Part A: from Day -1 (admission) to Day 12 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: Liters/hour (L/h)
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 9 | 9
Liters/hour (L/h) | 2.132 [1.16 to 4.06] | 3.232 [2.34 to 5.37]

16. Primary Outcome: Apparent Oral Clearance (CL/F) of Pamiparib in Plasma for Part B
Time Frame: Part B: from Day -1 (admission) to Day 9 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: Liters/hour (L/h)
Arm/Group | Part B: Pamiparib | Part B:Pamiparib + Itraconazole
Number analyzed (Participants) | 11 | 9
Liters/hour (L/h) | 1.987 [0.78 to 10.94] | 2.147 [0.86 to 12.97]

17. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Pamiparib in Plasma for Part A
Time Frame: Part A: from Day -1 (admission) to Day 12 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: Liters
Arm/Group | Part A: Pamiparib | Part A: Pamiparib + Rifampin
Number analyzed (Participants) | 9 | 9
Liters | 35.491 [22.61 to 51.12] | 37.712 [29.88 to 53.98]

18. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE is defined as any AE with an onset date on or after the date of first dose of study medication until the date of last study medication dose plus 30 days. Seriousness of the AE is determined by the investigator based on seriousness criteria.
Time Frame: From the date informed consent has been signed until last study medication dose plus 30 days (up to approximately 26 months)
Population: Safety Analysis Set includes all participants who received at least 1 dose of pamiparib
Measure: Number; unit: Number of participants
Groups:
- Core Phase: Arm B: Pamiparib + Itraconazole: Participants received 20 mg pamiparib orally from Days 1 and 7 fasting at least 8 hours pre-dose + 200 mg itraconazole orally 30 minutes after meal Day 3 to Day 8
Arm/Group | Core Phase: Arm A: Pamiparib + Rifampin | Core Phase: Arm B: Pamiparib + Itraconazole | Extension Phase
Number analyzed (Participants) | 12 | 13 | 24
Number of participants
  All TEAEs | 5 | 6 | 18
  Serious TEAEs | 0 | 1 | 2

19. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Assessments, Vital Signs, ECG Parameters and Physical Examinations
Time Frame: Up to approximately 26 months
Population: Safety Population
Measure: Number; unit: Number of participants
Arm/Group | Core Phase: Arm A: Pamiparib + Rifampin | Core Phase: Arm B: Pamiparib + Itraconazole | Extension Phase
Number analyzed (Participants) | 12 | 13 | 24
Number of participants
  Laboratory Assessments | 0 | 0 | 0
  Vital Signs | 0 | 0 | 0
  Physical Examinations | 0 | 0 | 0
  ECG Parameters | 0 | 0 | 0

20. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Pamiparib in Plasma for Part B
Time Frame: Part B: from Day -1 (admission) to Day 9 (discharge); 30 min pre-dose, 0.5, 1, 2, 4, 6, 9, 12 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: Liters
Arm/Group | Part B: Pamiparib | Part B:Pamiparib + Itraconazole
Number analyzed (Participants) | 12 | 12
Liters | 34.697 [21.60 to 70.69] | 37.589 [24.21 to 69.03]

ADVERSE EVENTS:
Time Frame: From the date informed consent has been signed until last study medication dose plus 30 days (up to approximately 26 months)
Arm/Group | Core Phase: Arm A: Pamiparib + Rifampin | Core Phase: Arm B: Pamiparib + Itraconazole | Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/13 | 2/24
Other Adverse Events (participants affected / at risk) | 5/12 | 6/13 | 18/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Arm A: Pamiparib + Rifampin (N=12) | Core Phase: Arm B: Pamiparib + Itraconazole (N=13) | Extension Phase (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Arm A: Pamiparib + Rifampin (N=12) | Core Phase: Arm B: Pamiparib + Itraconazole (N=13) | Extension Phase (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 11 (15)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenogastric reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (5)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT03994211/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03994211/SAP_001.pdf